CLINICAL TRIAL: NCT03373175
Title: Influence of Ventilator Model and Pressure Support Level in Muscular Unloading in COPD Patients With Non Invasive Ventilation (NIV)
Brief Title: Assesment of Muscular Unloading in Chronic Obstructive Pulmonary Disease (COPD) Patients With NIV
Acronym: EMGNIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Manel Lujan-Torne, MD, Corporacion Parc Tauli
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017632
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: COPD
Keywords: Monitoring NIV, inspiratory muscular unloading, EMG
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ventilator 1 vs Ventilator 2 (Experimental): 2 Ventilators will be evaluated for patient. All parameters will be monitored and the differences will be analyzed. Interventions: Basal record Pressure Support 10 (PS 10)record Pressure Support 15 (PS 15) record Pressure Support 20 (PS 20) record
  Interventions: Device: Basal record; Device: PS 10 record; Device: PS 15 record; Device: PS 20 record
- Ventilator 3 vs Ventilator 4 (Experimental): 2 Ventilators will be evaluated for patient. All parameters will be monitored and the differences will be analyzed.Interventions: Basal record PS10 record PS15 record PS 20 record
  Interventions: Device: Basal record; Device: PS 10 record; Device: PS 15 record; Device: PS 20 record
- Ventilator 5 vs Ventilator 6 (Experimental): 2 Ventilators will be evaluated for patient. All parameters will be monitored and the differences will be analyzed. Interventions: Basal record PS10 record PS15 record PS 20 record
  Interventions: Device: Basal record; Device: PS 10 record; Device: PS 15 record; Device: PS 20 record
- Ventilator 7 vs Ventilator 8 (Experimental): 2 Ventilators will be evaluated for patient. All parameters will be monitored and the differences will be analyzed. Interventions: Basal record PS10 record PS15 record PS 20 record
  Interventions: Device: Basal record; Device: PS 10 record; Device: PS 15 record; Device: PS 20 record

INTERVENTIONS:
Device: Basal record — Basal EMG record will be performed during 5 minutes. This record must be the same in both ventilators.
Device: PS 10 record — PS 10 EMG record record will be performed during 5 minutes. First with ventilator 1 and then with the other. The patient must be rest at least 5 minutes to recover basal record
Device: PS 15 record — PS 15 EMG record record will be performed during 5 minutes. First with ventilator 1 and then with the other. The patient must be rest at least 5 minutes to recover basal record
Device: PS 20 record — PS 20 EMG record record will be performed during 5 minutes. First with ventilator 1 and then with the other. The patient must be rest at least 5 minutes to recover basal record

SUMMARY:
Evaluation of high intensity NIMV in terms of physiological parameters has been performed in short-term studies in COPD patients. However, the support pressure levels used in exacerbated patients seem contradictory and the muscular unloading levels are uncertain. The objective of study is to determine the discharge level of the inspiratory musculature reached at the same pressure support (PS) values in a group of hospital and domiciliary ventilators. Patients with COPD in at least 6 months of treatment with home NIMV and in stable phase of their disease will be included. Eight commercial ventilators will be used, each patient will use 2 different ventilators. A 5 minute record will be taken at baseline (without NIMV). Subsequently, 5 minutes in NIMV in 3 levels of PS (15/10/20) for each ventilator (15/10/20) and patient with expiratory positive airway pressure (EPAP) of 5 centimeters of water (cmH2O) will be recorded. The results will be compared between the different ventilators and PS values using a general linear model for repeated variables to determine the differences between ventilators and PS levels of respiratory muscular unloading in COPD patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD diagnoses based on a spirometry performed the previous year during stability.
* COPD patients with home NIV treatment of at least 6 months with acceptable compliance and adaptation.
* Stable patients or just before hospital discharge due to an exacerbation with gasometric stability.

Exclusion Criteria:

* Respiratory acidosis in blood gas analysis, just in case of recent exacerbation
* Patients with restrictive pathology and /or obesity (IMC>35)
* Poor quality of EMG signals.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscular unloading (µv) | 1 day
  Differences in parasternal electromyogram (EMG) signals interpretation between the record of ventilator 1 and ventilator 2.

SECONDARY OUTCOMES:
Baseline EMG (µv) record | 1 day
  Parasternal EMG signals interpretation before and without NIV. Spontaneous breathing record. The outcome measure inspiratory muscular effort of the patient in basal conditions.
Pressure support 10 EMG (µv) record. V1 | 1 day
  Parasternal EMG signals interpretation during first phase of NIV, in this case it will be programmed at 10 cmH2O os pressure support (PS) with Ventilator 1 during 5 minutes.
Pressure support 15 EMG (µv) record. V1 | 1 day
  Parasternal EMG signals interpretation during the second phase of NIV that will be programmed at 15 cmH2O os pressure support (PS) with Ventilator 1 during 5 minutes
Pressure support 20 EMG (µv) record. V1 | 1 day
  Parasternal EMG signals interpretation during the last phase of NIV that will be programmed at 20 cmH2O os pressure support (PS) with Ventilator 1 during 5 minutes
Pressure support 10 EMG (µv) record. V2 | 1 day
  Paraesternal EMG signals interpretation during the last phase of NIV that will be programmed at 10 cmH2O os pressure support (PS) with Ventilator 2 during 5 minutes
Pressure support 15 EMG (µv) record. V2 | 1 day
  Parasternal EMG signals interpretation during the last phase of NIV that will be programmed at 15 cmH2O os pressure support (PS) with Ventilator 2 during 5 minutes
Pressure support 20 EMG (µv) record. V2 | 1 day
  Parasternal EMG signals interpretation during the last phase of NIV that will be programmed at 20 cmH2O os pressure support (PS) with Ventilator 2 during 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Manel Lujan, MD, Principal Investigator — Corporacion Parc Tauli (Sabadell, Barcelona); Javier Sayas, Principal Investigator — Hospital Universitario 12 de Octubre (Madrid)
Locations (2):
- Spain (2):
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Derived] Lalmolda C, Florez P, Corral M, Hernandez Voth A, Grimau C, Sayas J, Lujan M. Does the Efficacy of High Intensity Ventilation in Stable COPD Depend on the Ventilator Model? A Bench-to-Bedside Study. Int J Chron Obstruct Pulmon Dis. 2022 Jan 14;17:155-164. doi: 10.2147/COPD.S327994. eCollection 2022. PMID 35058690